CLINICAL TRIAL: NCT02930928
Title: Evaluation of an Algorithm for Gender Specific and Habitus Adapted Length Based Body Weight Estimation in Children - Improvement by Adding Another Parameter?
Brief Title: Can Habitus Adapted Length Based Body Weight Estimation be Improved by Adding Further Parameters?
Acronym: Including MUC
Status: Completed | Type: Observational
Sponsor: University Children's Hospital, Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: KEK-ZH-Nr. 2015-0191 - Part 4
Record Dates: First submitted 2016-10-10; First posted 2016-10-12 (Estimated); Last update posted 2020-11-10 (Actual); Status verified 2020-11

CONDITIONS: Weight-Estimation
Keywords: Anaesthesia; Anthropometry; Body weight and measures; Development; Emergency treatment; Patient safety
MeSH Terms: conditions — Body Weight

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Accuracy of weight estimation: Computer based comparison of the two algorithms based on collected patient data
  Interventions: Other: Accuracy of weight estimation

INTERVENTIONS:
Other: Accuracy of weight estimation — Computer based comparison

SUMMARY:
The purpose of this prospective single center study is to investigate if the accuracy of length based body weight estimation by the already investigated algorithm (CLAWAR) can be improved by adding another parameter. For this study 500 patients are required to collect anonymized data (length, weight, age, mid upperarm circumference and patient habitus by visual estimation) for achieving a power of 80% during statistical analysis. The main hypothesis ist that CLAWAR's accuracy can be improved.

DETAILED DESCRIPTION:
This prospective single center study is performed at the university children's Hospital zurich. Patients planned for surgery in general anaesthesia with intubation, aged 0 to 16 years and with a body length suitable for CLAWAR. Patient and parental information is performed during the pre-anaesthetic visit.

After written consent the patient will be included. Patient ́s length and weight will be measures earliest one day before data collection. Data collection during anaesthesia has no influence on the daily anaesthesia routine and has no impact on patient safety and anaesthesia. Patient's data is made anonymous for further inspection. Data is documented in Microsoft Excel and statistical analysis calculated with SPSS.

500 patients are needed for a power of 80%. Primary outcome parameter is the accuracy of length based weight estimation using either patient habitus by visual estimation or an improved version of the algorithm CLAWAR using the mid upperarm circumference.

ELIGIBILITY:
Inclusion Criteria:

* body length suitable with the investigated algorithm
* all patients aged 0 -16 years

Exclusion Criteria:

* already included in this study once
* missing patient or parental consent

Ages: 1 Day to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Pediatric patients planned for elecitve surgery in general anaesthesia
Sampling Method: Probability Sample
Enrollment: 495 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
length-based weight-estimation by algorithm | during procedure
  Habitus adapted weight estimation based on visual habitus classification compared to weight estimation by the modified algorithm CLAWAR utilizing mid upperarm circumference

CONTACTS AND LOCATIONS:
Overall Officials: Alexander R Schmidt, MD, Principal Investigator — University Children's Hospital Zurich, Department of Anaesthesia
Locations (1):
- University Childrens Hospital, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No